CLINICAL TRIAL: NCT04813445
Title: Analysing the Effects of Xingnaojing for Mild-to-severe Acute Ischemic Stroke(AXAIS): A Multicenter, Randomized, Open-label, Controlled Trial
Brief Title: Analysing the Effects of Xingnaojing for Mild-to-severe Acute Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dongzhimen Hospital, Beijing (Other)
Collaborators: Affiliated Hospital of Nantong University (Other); Nanjing Brian Hospital (Other); Affiliated Hospital of Chengde Medical University (Other)
Responsible Party: Principal Investigator, Ying Gao, Principal Investigator, Clinical Professor, Dongzhimen Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018YFC1705001-05
Record Dates: First submitted 2021-03-16; First posted 2021-03-24 (Actual); Last update posted 2022-02-18 (Actual); Status verified 2022-02

CONDITIONS: Acute Stroke; Ischemic Stroke
MeSH Terms: conditions — Stroke; Ischemic Stroke | interventions — xingnaojing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Xingnaojing injection (Experimental): Subjects will receive intravenously administered Xingnaojing injection, combined with guidelines-based standard care.
  Interventions:
  Drug: Xingnaojing injection Other: Standard care
  Interventions: Drug: Xingnaojing injection
- Standard care (No Intervention): Subjects will receive guidelines-based standard care.
  Interventions:
  Other: Standard care

INTERVENTIONS:
Drug: Xingnaojing injection — Xingnaojing injection (20 ml)+0.9% diluted sodium chloride injection 250ml, IV (in the vein), every 12 hours for 10 days.
  Arms: Xingnaojing injection

SUMMARY:
The main purpose of this trial is to analyse the Effects of Xingnaojing for Mild-to-severe Acute Ischemic Stroke by Metabonomics, proteomics and clinical parameters.

DETAILED DESCRIPTION:
Xingnaojing is widely used in China, but there is lack of sufficient and reasonable explanation of its intervention effects for acute ischemic stroke currently. The primary hypothesis of this trial is that , Compared with the blank control group, Xingnaojing will produce serial changes in plasma and urine metabolites and biomarkers at baseline (pre-dose), 8 days and 11days . The serial changes may be the potential support to explain the intervention effect of Xingnaojing. All participants will have a National Institutes of Health Stroke Scale(NIHSS)entry score of 4-25. Participants who have planned or already received the intravenous thrombolysis or endovascular treatment will be excluded. The primary outcome will be determined at 11 days.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute ischemic stroke；
* Symptom onset within 24 hours；
* 35 ≤ Age ≤ 80 years；
* 4 ≤ NIHSS ≤ 25；
* Patient or legally authorized representative has signed informed consent.

Exclusion Criteria:

* Expected length of hospital stay is less than 10 days;
* Planned or already receiving intravenous thrombolysis or endovascular treatment;
* Use of drugs with unknown composition within 1 week before enrollment;
* Patients with acute infectious diseases (e.g. acute pneumonia) or taking related drugs within 1 month before treatment in the group;
* Suspected secondary stroke caused by tumor, brain trauma, or hematological diseases;
* Already dependent in activities of daily living before the present acute stroke (defined as modified Rankin Scale score ≥ 2) ;
* Other conditions that cause cardiogenic embolism (e.g., atrial fibrillation, rheumatic heart disease, valvular heart disease);
* Other conditions that lead to motor dysfunction (e.g., severe osteoarthrosis, rheumatoid arthritis);
* Significant renal or hepatic insufficiency (defined as a serum creatinine concentration, alanine aminotransferase (ALT), or aspartate aminotransferase (AST) value that is twice the upper limit of normal);
* Life expectancy of 3 months or less due to other life-threatening illness (e.g.,advanced cancer)
* Other conditions that render outcomes or follow-up unlikely to be assessed;
* Known to be pregnant or breastfeeding;
* Currently receiving an investigational drug.

Ages: 35 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2021-05-28 (Actual); Primary Completion 2022-06-28 (Estimated); Study Completion 2022-09-28 (Estimated)

PRIMARY OUTCOMES:
The change of NIHSS score | Baseline, 3 days, 7 days and 10 days
  The NIHSS score ranges from 0 (best score) to 42 (worst score).

SECONDARY OUTCOMES:
The proportion of NIHSS score from 0 to 1 | Baseline, 3 days, 7 days and 10 days
  The NIHSS score ranges from 0 (best score) to 42 (worst score).
Patient reported outcome (PRO) scale of stroke | 10 days
  Patient reported outcome (PRO) scale of stroke at 10 days.The PRO score ranges from 0(worst score) to 180 (best score).
The proportion of patients independent at 30 days and 90 days | 30 days and 90 days
  The proportion of patients independent is defined as Modified Rankin Scale score of 0, 1, or 2. The mRS score ranges from 0 (best score) to 6 (worst score).
Cardio-cerebral vascular incident | Within baseline and 90 days
  Cardio-cerebral vascular incident were defined as stroke, acute coronary syndrome (acute ST-elevation myocardial infarction, acute non-ST-elevation myocardial infarction and unstable angina), vascular death, etc.
The difference in proteomic and metabolomics | baseline (pre-dose), 7 days and 11days
  Through proteomics and metabonomics to explore whether there are different metabolites or proteins between the two groups.（It's not known whether there are differences in the human body between the two groups.We are in the exploratory stage.）
State of consciousness | Baseline, 3 days, 7 days and 10 days
  The state of consciousness evaluated by Glasgow Coma Scale at Baseline, 3 days, 7 days and 10 days. The Glasgow score ranges from 3(worst score) to 15 (best score).
Activities of daily living | 30 days and 90 days
  Activities of daily living will be measured by Barthel Index score at 30 days and 90 days.The Barthel Index score ranges from 0 (worst score) to 100 (best score).
Safety end points | 10 days
  Number of patients with any adverse events, results of electrocardiography, vital signs and laboratory tests (complete blood count, chemistry and urinalysis).
Stroke related deaths and deaths from any cause | Within 10 days and 90 days
  Stroke related deaths and deaths from any cause within 10 days and 90 days after symptom onset.

CONTACTS AND LOCATIONS:
Locations (1):
- Dongzhimen Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No